CLINICAL TRIAL: NCT06710496
Title: HISTOLOGICAL RESULTS IN TRANSGENDER INDIVIDUALS ASSIGNED TO FEMALES AT BIRTH UNDERGOING GENDER AFFIRMATION SURGERY AND IN TESTOSTERONE THERAPY
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Maria Cristina Meriggiola, Professor Maria Cristina Meriggiola, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: ISTO-AFAB
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-09

CONDITIONS: Pregnancy; Smoking Behavior; Testosterone Replacement Therapy; Drugs; Comorbidities and Coexisting Conditions; Gynecological Surgery; Transgender Men; Gender Affirmation Surgery; Hormone Replacement Therapy; Gynecological Disorders
Keywords: transgender; afab; histology
MeSH Terms: conditions — Smoking; Genital Diseases, Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AFAB TG: assigned female at birth transgender people undergoing gender affirming surgery during testosterone therapy
  Interventions: Other: analysis of medical records

INTERVENTIONS:
Other: analysis of medical records — analysis of medical records of the patients

SUMMARY:
The aim of this study is to report histological results of genital organs removed during gender affirmg surgery in transgender people assigned female at birth (AFAB), to increase the knowledge about the long-term effects of gender affirming hormone therapy with testosterone on these organs and to evaluate the incidence of benign and malign gynecological pathology in AFAB transgender people.

DETAILED DESCRIPTION:
This retrospective, observational, single-center study aims to analyze histological data obtained from the analysis of ovaries, fallopian tubes, uterine body, endometrium, and cervix of assigned female at birth (AFAB) transgender individuals who underwent gender affirming surgey (GAS) with hysterectomy and bilateral adnexectomy or hysterectomy alone following the administration of exogenous Testosterone (T). Histological results of the genital organs removed during GAS can provide important information about the effects and safety of loong term T treatment on these organs. Data on this subject is scarce in the literature. For this reason, even today, pathologists have not been able to establish guidelines for describing the histological results obtained from these patients.Furthermore, this analysis will evaluate the incidence of benign and malignant gynecological pathology in AFAB transgender people.

ELIGIBILITY:
Inclusion Criteria:

* gender incongruence diagnosis
* people assigned female at birth
* age >18 years
* gender affirming surgery with hysterectomy
* testosterone therapy

Exclusion Criteria:

* previous gynecological surgery
* previous gynecological disorder diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: transgender people assigned female at birth undergoing gender affirming surgery with hysterectomy and on testosterone therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
histological description of genital organs | 6 months

SECONDARY OUTCOMES:
prevalence of malignant and benign gynecological pathology | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- irccs azienda ospedaliero universitaria di Bologna, Bologna, Emilia-Romagna, Italy